CLINICAL TRIAL: NCT02712268
Title: Intervention to Improve Appropriate Prescribing and Reduce Polypharmacy in Elderly Patients Admitted to an Internal Medicine Unit
Brief Title: Intervention to Improve Prescribing in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/039
Record Dates: First submitted 2016-02-29; First posted 2016-03-18 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Elderly Internal Medicine Patients
Keywords: Polypharmacy; Clinical decision-making
MeSH Terms: interventions — Checklist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- After introduction of the checklist (Other): Review of medications of all consecutive admitted patients during the study period using a checklist
  Interventions: Other: Checklist

INTERVENTIONS:
Other: Checklist — Introduction of a 5-point checklist to be used by all physicians on the internal medicine wards to review and adapt the medications of the patient.

SUMMARY:
This study tested the efficacy of an easy-to-use checklist aimed at supporting the therapeutic reasoning of physicians in order to reduce inappropriate prescribing and polypharmacy in elderly adults admitted to an internal medicine unit.

DETAILED DESCRIPTION:
Background: Polypharmacy and inappropriate medication prescriptions are associated with increased morbidity and mortality. Most interventions proposed to improve appropriate prescribing are time and resource intensive and therefore hardly applicable in daily clinical practice.

Objective: To test the efficacy of an easy-to-use checklist aimed at supporting the therapeutic reasoning of physicians in order to reduce inappropriate prescribing and polypharmacy.

Design: single-center, interventional, quasi-experimental before-after study. Patients: Consecutive patients aged ≥65 years, hospitalized in the division of internal medicine of a Swiss secondary-level hospital from September to November 2012 (control group, N=450) and from September to November 2013 (intervention group, N=450).

Intervention: Introduction of a 5-point checklist to be used by all physicians on the internal medicine wards.

Main Measures: The proportion of patients with prescription of potentially inappropriate medications (PIMs) at discharge, according to Screening tool of older people's prescriptions (STOPP) criteria, and the number of prescribed medications at discharge, before and after the introduction of the checklist. Secondary outcomes were the prevalence of polypharmacy (≥ 5 drugs) and hyperpolypharmacy (≥ 10 drugs), and the prevalence of potentially inappropriate prescribing omissions (PPOs) according to START criteria.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged ≥65 years,
* patients hospitalized in the division of internal medicine of a Swiss secondary-level hospital from September to November 2012 (control group, N=450) and from September to November 2013 (intervention group, N=450).

Exclusion Criteria:

* none

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 450 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of patients prescribed potentially inappropriate medications (PIM) at discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  The proportion of patients prescribed PIMs at discharge, according to STOPP (Screening Tool of Older Person's potentially inappropriate Prescriptions) criteria, before and after the introduction of the checklist.
Change in the number of prescribed medications at discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  Number of prescribed medications at discharge, before and after the introduction of the checklist.

SECONDARY OUTCOMES:
Number of prescribed drugs at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
Prevalence of polypharmacy at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  concomitant use of more than 5 drugs
Prevalence of hyperpolypharmacy at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  concomitant use of more than 10 drugs
Prevalence of potentially inappropriate prescribing omissions (PPO) at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  according to START (Screening Tool of Alert doctors to the Right Treatment) criteria
Number of patients prescribed NSAID at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  Non-steroidal anti-inflammatory drugs (NSAID)
Rate (%) of inappropriate prescriptions of NSAID at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  Non-steroidal anti-inflammatory drugs (NSAID)
Number of patients prescribed proton pump inhibitors at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  proton pump inhibitor (PPI)
Rate (%) of inappropriate prescriptions of proton pump inhibitors at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  proton pump inhibitor (PPI)
Number of patients prescribed systemic corticosteroids at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
Rate (%) of inappropriate prescriptions of systemic corticosteroids at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
Number of patients prescribed metamizole at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
Rate (%) of inappropriate prescriptions of metamizole at admission and discharge | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
In-Hospital mortality rate | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
All-cause re-hospitalization rate | In the 3 months after introduction of the checklist (Sept.-Nov. 2013, intervention group) and in 3 months (Sept.-Nov. 2012) one year before the introduction of the checklist (control group)
  re-hospitalization rate 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bassetti, MD, Principal Investigator — University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data are available.